CLINICAL TRIAL: NCT00685672
Title: Pharmacokinetic Interaction Effects of Combined Fentanyl and Adrenalin in Epidural Analgesia During Child Birth
Brief Title: Safety of Epidural Fentanyl and Adrenalin During Childbirth
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: edaadr-07; EUDRACT 2007-000322-52
Record Dates: First submitted 2008-05-21; First posted 2008-05-28 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy; Pain
Keywords: labor analgesia; fentanyl; epinephrine
MeSH Terms: conditions — Pain | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): adrenalin
  Interventions: Drug: adrenalin
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: adrenalin — adrenalin 2 microgram pr ml placebo
  Arms: 1
Drug: placebo — Saline instead of adrenaline in the epidural mixture
  Arms: 2

SUMMARY:
Investigation of pharmacokinetic effects of combining fentanyl and adrenalin in the epidural solution given to women in childbirth

DETAILED DESCRIPTION:
Healthy women with indication for labor epidural at the Labor Clinic, Rikshospitalet University Hospital, may be included. A randomized, placebocontrolled, double blind,comparison of epidural with and without adrenalin. Outcome: Length of birth, quality of pain relief, total amount of epidural solution injected, and plasma concentration of fentanyl.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at term in active labor

Exclusion Criteria:

* age below 18 years
* BMI > 40
* drug hypersensitivity

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of fentanyl | hours

SECONDARY OUTCOMES:
length of active labor | hours

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Dahl, PhD MD, Study Director — Dep of Anesethesiology, Akershus University Hospital
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lørenskog
  - Division of Anaesthesiology and Intensive Care Medicine, Rikshospitalet University Hospital, Oslo

REFERENCES:
- [Derived] Haidl F, Rosseland LA, Spigset O, Dahl V. Effects of Adrenaline on maternal and fetal fentanyl absorption in epidural analgesia: A randomized trial. Acta Anaesthesiol Scand. 2018 Oct;62(9):1267-1273. doi: 10.1111/aas.13175. Epub 2018 Jun 25. PMID 29943508